CLINICAL TRIAL: NCT03380416
Title: Medium-term Effects of a Portfolio Diet on Non-alcoholic Fatty Liver Disease in Type 2 Diabetic Patients
Brief Title: Effects of a Portfolio Diet on NAFLD in Type 2 Diabetic Patients
Acronym: MEDEA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, rivellese angela, Full Professor, Federico II University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16/17
Record Dates: First submitted 2017-10-30; First posted 2017-12-21 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2020-03

CONDITIONS: Diabetes Type 2; NAFLD
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Portfolio Diet (Experimental): The participants will follow a weight-maintaining diet characterized by whole-grain, polyphenol-rich foods, omega 3- rich foods, MUFA-rich foods (protein 18%/total energy, carbohydrates 41%/total energy, fat 41%/total energy, MUFA 26%/total energy, fiber 24 g/1000Kcal) polyphenols 2715/day, omega-3 2.6 g/day and omega-6 9.6 g/day)
  Interventions: Other: Portfolio Diet
- MUFA Diet (Active Comparator): The participants will follow a weight-maintaining diet characterized by MUFA-rich food (olive oil) (protein 18%/total energy, carbohydrates 41%/total energy, fat 41%/total energy, MUFA 28%/total energy, fiber 10 g/1000Kcal) polyphenols 376/day, omega-3 1.1 g/day and omega-6 7.4 g/day)
  Interventions: Other: MUFA Diet

INTERVENTIONS:
Other: Portfolio Diet — Medium-term (8 weeks ) nutritional intervention
  Arms: Portfolio Diet
Other: MUFA Diet — Medium-term (8 weeks ) nutritional intervention used as control
  Arms: MUFA Diet

SUMMARY:
Patients with type 2 diabetes and non-alcoholic fatty liver disease will be enrolled.

According to a parallel design, the participants will be randomized to a Portfolio diet or a monounsaturated fatty acid (MUFA)-rich diet (used as control) for 8 weeks.

At the beginning and at the end of the trial, the participants will undergo a MRI spectroscopy to evaluate fatty liver content. Moreover, the participants will undergo a test meal resembling the nutritional composition of the assigned diet to evaluate fasting and postprandial metabolic response.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes
* non-alcoholic fatty liver disease (evaluated by US)
* HbA1c <7.5%
* LDL cholesterol <130 mg/dl

Exclusion Criteria:

* hypoglycemic therapy with sodium-glucose cotransporter (SGLT-2), pioglitazone and glucagon-like peptide (GLP-1) analogues
* severe liver and kidney failure
* recent cardiovascular events (prior 6 months)
* any other acute/chronic disease (anemia, cancer, BPCO)

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2017-04-04 (Actual); Primary Completion 2019-03-07 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
Liver fat content | Change from Baseline after 8 weeks
  MRI spectroscopy

SECONDARY OUTCOMES:
Liver functionality | Change from Baseline after 8 weeks
  Liver enzymes
Blood pressure | Change from Baseline after 8 weeks
Endothelial function | Change from Baseline after 8 weeks
  Flow-mediated dilation
Liver fibrosis | Change from Baseline after 8 weeks
  Transient Elastography
Biochemical parameters | Change from Baseline after 8 weeks
  glucose homeostasis (glucose)
Body composition | Change from Baseline after 8 weeks
  bioimpedance analyses (BIA)
lipids | Change from Baseline after 8 weeks
subclinical inflammation | Change from Baseline after 8 weeks
  elisa
oxidative stress | Change from Baseline after 8 weeks
  urinary isoprostanes
Biochemical parameters | Change from Baseline after 8 weeks
  glucose homeostasis (HbA1c)
Biochemical parameters | Change from Baseline after 8 weeks
  glucose homeostasis (Insulin)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Clinical Medicine and Surgery, Naples, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Costabile G, Salamone D, Della Pepa G, Testa R, Vitale M, Brancato V, Salvatore M, Soricelli A, Annuzzi G, Rivellese AA, Bozzetto L. ApoC-III and ectopic fat accumulation in individuals with type 2 diabetes: an exploratory analysis from the MEDEA randomised controlled study. Diabetologia. 2025 Sep;68(9):2036-2041. doi: 10.1007/s00125-025-06464-w. Epub 2025 Jun 5. PMID 40471240
- [Derived] Della Pepa G, Brancato V, Costabile G, Salamone D, Corrado A, Vitale M, Cavaliere C, Mancini M, Salvatore M, Luongo D, Riccardi G, Rivellese AA, Annuzzi G, Bozzetto L. An Isoenergetic Multifactorial Diet Reduces Pancreatic Fat and Increases Postprandial Insulin Response in Patients With Type 2 Diabetes: A Randomized Controlled Trial. Diabetes Care. 2022 Sep 1;45(9):1935-1942. doi: 10.2337/dc22-0605. PMID 35862001
- [Derived] Costabile G, Della Pepa G, Salamone D, Luongo D, Naviglio D, Brancato V, Cavaliere C, Salvatore M, Cipriano P, Vitale M, Corrado A, Rivellese AA, Annuzzi G, Bozzetto L. Reduction of De Novo Lipogenesis Mediates Beneficial Effects of Isoenergetic Diets on Fatty Liver: Mechanistic Insights from the MEDEA Randomized Clinical Trial. Nutrients. 2022 May 23;14(10):2178. doi: 10.3390/nu14102178. PMID 35631319
- [Derived] Della Pepa G, Vetrani C, Brancato V, Vitale M, Monti S, Annuzzi G, Lombardi G, Izzo A, Tommasone M, Cipriano P, Clemente G, Mirabelli P, Mancini M, Salvatore M, Riccardi G, Rivellese AA, Bozzetto L. Effects of a multifactorial ecosustainable isocaloric diet on liver fat in patients with type 2 diabetes: randomized clinical trial. BMJ Open Diabetes Res Care. 2020 May;8(1):e001342. doi: 10.1136/bmjdrc-2020-001342. PMID 32448788